CLINICAL TRIAL: NCT05458622
Title: 3TR (Taxonomy, Treatment, Targets and Remission) Systemic Lupus Erithematosus Study Protocol
Acronym: 3TR-SLE1
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 29BRC21.0367 (3TR-SLE1)
Record Dates: First submitted 2022-06-13; First posted 2022-07-14 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Systemic Lupus Erythematosus (SLE)
Keywords: Systemic; Lupus; Erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — Blood Specimen Collection; Histocompatibility Testing

STUDY DESIGN:
Intervention Model Description: Patients with stable or quiescent SLE will be included and followed-up in routine clinical care until a flare or until the 2 years end-of-study (EOS) visit.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Stable or quiescent SLE (Other): Patients included in this study will undergo one assessment at the time of recruitment and at the time of the end of study (time of a flare or at least 24 months after inclusion)
  The following information will be collected :
  * General data: date of flare.
  * Disease activity: BILAG; SLEDAI-2K; PhGA (0-3); PGA (0-10); LLDAS; DORIS ; CLASI for mucocutaneous involvement; 44 joint assessment; proteinuria (UPCR); serum creatinine and eGFR for lupus nephritis.
  * Organ damage: SLICC/ACR Damage Index.
  * Kidney histopathology
  * HRQoL: EQ-5D-5L; FACIT-F; Medical Outcomes Study 36-item Short Form health survey (SF-36); Epworth Sleepiness scale (ESS); Lupus-QoL.
  * Start day and current dose for current treatments
  Biological samples which will be obtained twice, at baseline and at the time of the first flare documented over 24 months, or at month 24 if no flare has been documented:
  * Blood
  * Urine
  * Stool
  * Saliva
  * Tissue samples for organ-specific manifestations
  Interventions: Biological: Blood sample; Biological: Urine sample; Biological: Saliva sample; Biological: Stood sample; Procedure: Tissue sample

INTERVENTIONS:
Biological: Blood sample — - Total volume of blood (on each sampling occasion): 54,5mL.
  * Whole blood will be collected in EDTA, 1 tube of 10 mL for DNA (genotyping, methylation arrays; at baseline for genotyping and at EOS visit for methylation arrays). From this, an aliquot of 0.5 mL for baseline cell numbers (cell proportions, CyTOF/flow cytometry) at all time points; capture of leukocytes for blood single cell RNA seq. at all time points and 5 mL for cell stimulations for cell metabolome (C13 to be added), and 1 tube of 10 mL for cell stimulations (CyTOF) at baseline.Tempus tube: 1 tube of 3 mL for RNA, 1 tube of 3mL for whole blood RNA seq.; to be taken at all time points. Plasma will be obtained and aliquoted from these tubes; to be obtained at all time points.
  * Serum: 2 tubes of 10 mL without anticoagulant for measurements of anti-drug antibodies, hydroxychloroquine levels, cytokines and analytes, proteome, and autoantibodies; to be taken at all time points.
Biological: Urine sample — - Urine: 100 mL which will be centrifuged. The pellet will be frozen, and the urine supernatant will be aliquoted;
Biological: Saliva sample — - Saliva: will be collect in special container for saliva microbiome and methylation;
Biological: Stood sample — - Stool: One sample for microbiome to be sent to the biobank, frozen at -80 °C
Procedure: Tissue sample — - Tissue samples for organ-specific manifestations:
  * Kidney tissue in lupus nephritis: one small fragment of the fresh kidney biopsy will be stored in a 10% dimethyl sulfoxide (DMSO) solution (slow freezing to -80 °C) until shipment.
  * Skin tissue (at selected centers) from inflamed lesion and non-inflamed skin from the gluteal region will be obtained through punch biopsy and stored in a 10% dimethyl sulfoxide (DMSO) solution (slow freezing to -80 °C) until shipment.
  * Synovial tissue (at selected centers) will be obtained through ultrasound-directed arthroscopy and stored in a 10% dimethyl sulfoxide (DMSO) solution (slow freezing to -80 °C) until shipment.
  * Aspirate from swollen lymph nodes (at selected centers) will be obtained and stored in a 10% dimethyl sulfoxide (DMSO) solution (slow freezing to -80 °C) until shipment.

SUMMARY:
The natural history of Systemic lupus erythematosus (SLE) is characterized by relapses or flares alternated with periods of remission. Flares are associated with accrual of organ damage independently of other risk factors, both contributing to a considerable morbidity. No useful biomarker is currently available to predict which patients with a quiescent disease are at risk of flare.

The 3TR project (funded by the Innovative Medicines Initiative 2 Joint Undertaking under grant agreement No 831434, and supported by European Union's Horizon 2020 research and innovation programme and EFPIA) is a transdisciplinary consortium that primary aims at identifying biosignatures as predictors of response and non-response to therapy in seven different autoimmune, allergic and inflammatory diseases, including SLE. 3TR will perform a longitudinal multi-dimensional molecular analysis in patients with these diseases. A molecular profiling approach is a modern and innovative way to investigate and stratify heterogeneous diseases on the basis of their common biomolecular pathways. The main hypothesis of the 3TR project is that data obtained from multiomic analysis across the seven different diseases will identify shared biological pathways that better predict the response or non-response to therapy despite their differences in terms of clinical phenotypes and pathogenetic mechanisms. Therefore patients from multiple European centers participating in 3TR will be recruited for a longitudinal clinical follow-up and collections of several samples that will be used to perform multi-omic analysis.

DETAILED DESCRIPTION:
The study will be carried out in the framework of the IMI2 (innovative medicine initiative) and EFPIA (European Federation of Pharmaceutical Industries and Associations)-funded 3TR (Taxonomy, Treatment, Targets and Remission) project. The programme is supported by the European Union's Horizon 2020 research and innovation programme. 3TR is funded under the grant agreement No 831434 and it runs from 2019 to 2026.

3TR is a transdisciplinary consortium that aims to perform a longitudinal multi-dimensional molecular analysis in patients with autoimmune, allergic and inflammatory diseases. A molecular profiling approach is a modern and innovative way to investigate and stratify heterogeneous diseases on the basis of their common biomolecular pathways. The main hypothesis of the 3TR project is that data obtained from multiomic analysis across seven different diseases, including SLE, will identify shared biological pathways that better predict the response or non-response to therapy despite their differences in terms of clinical phenotypes and pathogenetic mechanisms. Patients from multiple European centers participating in 3TR will be recruited for a longitudinal clinical follow-up and collections of several samples that will be used to perform multi-omic analysis.

Several innovations are expected within the 3TR project to increase the knowledge of pathogenetic mechanisms underlying the clinical phenotypes in SLE, and to unravel, in the complexity of SLE biomolecular heterogeneity, the pathways of response or non-response to treatment, as well as, at an earlier stage, the processes that may lead to disease flare. These insights could ultimately allow the possibility to effectively practice prevention and counselling, to adopt measures of personalized treatment or to perform drug repurposing using the knowledge gained from the SLE studies and the studies on other diseases within the 3TR project.

Moreover, the impact of the COVID-19 viral pandemic will be implemented in our research. More specifically, we will investigate the impact of the presence of anti-SARS-CoV-2 antibodies of different isotypes (IgA, IgG, IgM) on the development of flare, as well as on the response or non-response to immunomodulatory therapy.

To implement the strategy, a two-step research has been designed, and comprises:

1. The flare biomarker study (3TR SLE 1) is considered a "feeding" phase before the main part. Patients who meet the inclusion criteria for 3TR SLE 2 will be proposed to participate in the second study.
2. The response biomarker study (3TR SLE 2), which is a prospective study (main part).

The present protocol relates to the flare biomarker study (3TR SLE 1).

ELIGIBILITY:
Inclusion Criteria:

1. Age at the time of inclusion ≥ 18 years;
2. Able to consent and agree to participate to the study.
3. Diagnosis of SLE according to the EULAR/ACR criteria; BILAG C, D or E only;
4. No restriction regarding current or previous therapies, except for hydroxychloroquine (HCQ) or chloroquine treatment which should be administered unless contraindicated or documented intolerance in the past.

Exclusion Criteria:

1. Pregnancy and/or breastfeeding;
2. Initiation or intensification of immunosuppressive therapy or a prednisone equivalent dose of > 10 mg/day within 30 days prior to baseline;
3. Unable or unaware to participate to the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2022-11-29 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Flare patient proportion according to the BILAG index at 24 months | 24 months
  Number of patients developing a flare within 24 months of follow-up, defined as a new BILAG A or B in any clinical domain.

SECONDARY OUTCOMES:
Proportion of flare according to the SELENA-SLEDAI Flare Index | Flare or 24 months
  Number of patients with a flare within 24 months, according to the SELENA-SLEDAI Flare Index (SFI). Flare will be defined as a 4-point increase in SLEDAI-2 K.
Anti-SARS-CoV-2 antibodies impact on risk of flare | Flare or 24 months
  Number of patients with anti-SARS-CoV-2 antibodies of different isotypes (IgA, IgG, IgM) with and without a flare during 24 months of follow-up.

CONTACTS AND LOCATIONS:
Locations (1):
- 01- CHU Brest, Brest, France

IPD SHARING:
Plan to Share IPD: Undecided